CLINICAL TRIAL: NCT03655262
Title: Treating Phobia With Multivoxel Neuro-reinforcement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Michelle Craske, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R61MH113772 (NIH)
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Results first posted 2023-12-27 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Phobia
Keywords: unconscious fear extinction; anxiety disorders; decoded neuro-reinforcement
MeSH Terms: conditions — Phobic Disorders; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 Session (Experimental): 1 neuro-reinforcement session
  Interventions: Behavioral: Unconscious Neuro-reinforcement
- 3 Sessions (Experimental): 3 neuro-reinforcement sessions
  Interventions: Behavioral: Unconscious Neuro-reinforcement
- 5 sessions (Experimental): 5 neuro-reinforcement sessions
  Interventions: Behavioral: Unconscious Neuro-reinforcement

INTERVENTIONS:
Behavioral: Unconscious Neuro-reinforcement — Individuals will complete an implicit fmri neuro-reinforcement task where real-time brain activity is matched to a desired activation. Individuals will also receive financial reward for activating the desired activation. Visual feedback will be presented to indicate how well individuals' brain activity matches the desired activation. Individuals will complete x day(s) of neuro-reinforcement.

SUMMARY:
Specific phobias and other anxiety disorders represent a major mental health problem, and present a significant challenge to researchers because effective treatment usually involves repeated exposure to feared stimuli, and the high levels of associated distress can lead to termination of treatment. Recent advances in computational functional magnetic resonance imaging (fMRI) provide a method by which individuals may be unconsciously exposed to fearful stimuli, leading to effective fear reduction while eliminating a primary cause of attrition.

The objective of the current study is to use the novel approach of neuro-reinforcement based on decoded fMRI information to reduce fear responses to fearful stimuli (e.g., spiders, heights) in individuals with phobias, directly and unconsciously in the brain, without repeatedly exposing participants to their feared stimuli.

Participants will be randomized into one of three groups of varying neuro-reinforcement sessions (1, 3, or 5). They will complete tests of subjective fear and directed attention while being scanned by fMRI to measure engagement of amygdala activity to fearful stimuli as well as measured through other indicators of fear such as skin conductance response.

DETAILED DESCRIPTION:
Anxiety disorders, the most common group of mental disorders in the United States, represent a major mental health problem. Phobias, in which fear and anxiety are triggered by a specific stimulus or situation, are the largest category of anxiety disorders and affect 5 - 12% of the world's population.

Exposure-based therapies are effective in reducing symptoms, but their effectiveness depends on the individual's capacity or willingness to consciously confront their feared object. The associated distress can be so extreme that it prevents patients from seeking treatment, and contributes to attrition from exposure once treatment begins. As a result, there is an unmet need for treatment that minimizes attrition and subjective patient discomfort.

The current study uses a novel technique of neuro-reinforcement based on decoded fMRI information to reduce fear responses to fearful stimuli directly and unconsciously without repeatedly exposing participants to those stimuli. The goals are to (1) confirm that our method decreases amygdala reactivity to images of phobic stimuli as well as (2) determine dosage-response optimization.

ELIGIBILITY:
Inclusion Criteria:

* Individual has normal or corrected to normal vision
* Individual has normal or corrected to normal hearing
* Individual is competent to understand informed consent

Exclusion Criteria:

* Individual is unable to fill in consent form correctly
* Individual is unable to respond adequately to screening questions
* Individual is unable to maintain focus or to sit during assessment
* Individual has history of: neurological disease or defect (e.g., stroke, traumatic brain injury, schizophrenia or other psychological disorders, or seizures)
* Individual has vision problems (including cataracts, amblyopia, or glaucoma)
* Individual presents with: PTSD, Obsessive Compulsive Disorder, Substance Use Disorder, Current Major Depression, Bipolar Disorder, Psychosis, neurologic diagnoses or unstable serious medical conditions
* Individual does not present with more than one object of specific phobia
* Individual can touch the phobic object category during the pre¬treatment Behavioral Approach Test without presenting significant distress
* Individual is currently prescribed psychotropic medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cushing CA, Lau H, Kawato M, Craske MG, Taschereau-Dumouchel V. A double-blind trial of decoded neurofeedback intervention for specific phobias. Psychiatry Clin Neurosci. 2024 Nov;78(11):678-686. doi: 10.1111/pcn.13726. Epub 2024 Sep 2. PMID 39221769
- [Derived] Cushing CA, Lau H, Kawato M, Craske MG, Taschereau-Dumouchel V. A double-blind trial of decoded neurofeedback intervention for specific phobias. medRxiv [Preprint]. 2024 Aug 1:2023.04.25.23289107. doi: 10.1101/2023.04.25.23289107. PMID 39132473

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1 Session | 3 Sessions | 5 Sessions
Started | 7 | 8 | 8
Completed | 7 | 8 | 7
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- 1 Session: 1 neuro-reinforcement session
  Unconscious Neuro-reinforcement: Individuals will complete an implicit fmri neuro-reinforcement task where real-time brain activity is matched to a desired activation. Individuals will also receive financial reward for activating the desired activation. Visual feedback will be presented to indicate how well individuals' brain activity matches the desired activation. Individuals will complete 1 day(s) of neuro-reinforcement.
- 3 Sessions: 3 neuro-reinforcement sessions
  Unconscious Neuro-reinforcement: Individuals will complete an implicit fmri neuro-reinforcement task where real-time brain activity is matched to a desired activation. Individuals will also receive financial reward for activating the desired activation. Visual feedback will be presented to indicate how well individuals' brain activity matches the desired activation. Individuals will complete 3 day(s) of neuro-reinforcement.
- 5 Sessions: 5 neuro-reinforcement sessions
  Unconscious Neuro-reinforcement: Individuals will complete an implicit fmri neuro-reinforcement task where real-time brain activity is matched to a desired activation. Individuals will also receive financial reward for activating the desired activation. Visual feedback will be presented to indicate how well individuals' brain activity matches the desired activation. Individuals will complete 5 day(s) of neuro-reinforcement.
- Total: Total of all reporting groups
Arm/Group | 1 Session | 3 Sessions | 5 Sessions | Total
Number analyzed (Participants) | 7 | 8 | 8 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 8 | 23
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26 (6.78) | 24.14 (14.24) | 25.86 (8.11) | 25.3 (9.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 4 | 18
  Male | 1 | 0 | 4 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 4 | 6
  Not Hispanic or Latino | 6 | 7 | 4 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 5 | 2 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 2 | 2 | 4 | 8
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Amygdala Reactivity
Description: The neural measure of difference in amygdala reactivity (measured by fMRI) to target phobic animals compared to control phobic animals from pre-treatment to post-treatment. Lower numbers (i.e. more negative numbers) indicate greater amygdala decrease and and better outcomes.
Time Frame: 10 days (measured at pre-treatment and post-treatment)
Measure: Mean (Standard Deviation); unit: Beta Coefficient
Arm/Group | 1 Session | 3 Sessions | 5 Sessions
Number analyzed (Participants) | 7 | 8 | 8
Beta Coefficient | -.691 (.796) | -.827 (1.620) | -.278 (1.682)

2. Primary Outcome: Subjective Fear Post-treatment Minus Pre-treatment
Description: Subjective Fear Ratings of images of targeted phobic stimuli
  Minimum score of 0, Maximum score of 180, higher scores mean worse outcome.
Time Frame: 10 days (measured at pre-treatment and post-treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 Session | 3 Sessions | 5 Sessions
Number analyzed (Participants) | 5 | 6 | 6
units on a scale | 0.32 (0.32) | -0.03 (0.37) | 0.43 (0.97)

3. Secondary Outcome: Skin Conductance Response: Physiological Arousal Post-treatment Minus Pre-treatment
Description: Skin conductance to image presentation of targeted phobic stimuli post-treatment minus pre-treatment
Time Frame: 10 days (measured at pre-treatment and post-treatment)
Measure: Mean (Standard Deviation); unit: Square Rooted Microsiemens
Arm/Group | 1 Session | 3 Sessions | 5 Sessions
Number analyzed (Participants) | 1 | 2 | 4
Square Rooted Microsiemens | -0.010 (0) | -0.097 (0.181) | -0.030 (0.192)

4. Secondary Outcome: Fear Survey Schedule
Description: Subjective fear ratings of a list of typical phobic stimuli
  Minimum score of 40, maximum of 200, higher scores mean worse outcome.
Time Frame: 10 days (measured at pre-treatment and post-treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 Session | 3 Sessions | 5 Sessions
Number analyzed (Participants) | 7 | 8 | 8
units on a scale | -2.46 (1.13) | -5.00 (1.12) | -11.93 (1.02)

5. Secondary Outcome: Stroop Task Post-treatment Minus Pre-treatment
Description: Measure of preferential allocation of attentional resources measured in reaction time (seconds) for visual presentation of the targeted phobic stimulus
Time Frame: 10 days (measured at pre-treatment and post-treatment)
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | 1 Session | 3 Sessions | 5 Sessions
Number analyzed (Participants) | 6 | 5 | 6
Seconds | -0.080 (.079) | -0.137 (.198) | -0.030 (.203)

ADVERSE EVENTS:
Time Frame: 2 years, 5 months
Arm/Group | 1 Session | 3 Sessions | 5 Sessions
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-23): https://cdn.clinicaltrials.gov/large-docs/62/NCT03655262/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-05): https://cdn.clinicaltrials.gov/large-docs/62/NCT03655262/SAP_001.pdf